CLINICAL TRIAL: NCT01816477
Title: A Prospective, Randomized, Controlled Trial of Post Operative Pain Control Using Ropivacaine and the ON-Q System in the Adult Pectus Excavatum Patient After Minimally Invasive Repair
Brief Title: Post Operative Pain Control Using Ropivacaine and the ON-Q System in the Adult Pectus Excavatum Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Halyard Health (Industry)
Responsible Party: Principal Investigator, Dawn E. Jaroszewski, Associate Professor of Surgery, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-008050
Record Dates: First submitted 2013-02-28; First posted 2013-03-22 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Pectus Excavatum
MeSH Terms: conditions — Funnel Chest | interventions — Injections, Epidural; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic epidural (Active Comparator): Thoracic epidural with Ropivicaine 0.25% placed pre-operatively by the anesthesiologist. Epidurals will remain in place for 72 hours and discontinued by the anesthesia pain management team.
  Interventions: Drug: Epidural (ropivicaine 0.25%)
- ON-Q soaker catheter system (Experimental): ON-Q soaker catheter system with Ropivicaine at 7 cc per hour placed by a single surgeon in the operating room. 7.5" catheters will be tunneled subcutaneously in the anterior axilla bilateral and secured with steri-strips and dressing. ON-Q systems will be primed with 750 cc and refilled accordingly to provide for 6 days of analgesia. Catheters will be removed by the surgeon in the hospital or clinic on the 6th post operative day. Patients may request removal of the catheter prior to the 6th day and this will not be considered a withdrawal from the study or complication and will be included in overall analysis, but noted accordingly.
  Interventions: Device: ON-Q soaker catheter system

INTERVENTIONS:
Device: ON-Q soaker catheter system — ON-Q soaker catheter system with Ropivicaine at 7 cc per hour placed by a single surgeon in the operating room. 7.5" catheters will be tunneled subcutaneously in the anterior axilla bilateral and secured with steri-strips and dressing. ON-Q systems will be primed with 750 cc and refilled accordingly to provide for 6 days of analgesia. Catheters will be removed by the surgeon in the hospital or clinic on the 6th post operative day. Patients may request removal of the catheter prior to the 6th day and this will not be considered a withdrawal from the study or complication and will be included in overall analysis, but noted accordingly.
  Arms: ON-Q soaker catheter system
Drug: Epidural (ropivicaine 0.25%) — Thoracic epidural with Ropivicaine 0.25% placed pre-operatively by the anesthesiologist. Epidurals will remain in place for 72 hours and discontinued by the anesthesia pain management team.
  Other Names: Naropin
  Arms: Thoracic epidural

SUMMARY:
Pectus excavatum (PE) is a common chest wall deformity where the sternum is displaced posteriorly. In severe cases, surgery is performed to correct the defect. In recent years, minimally invasive surgery with the placement of stainless steel support bars has been increasingly performed in patients over the age of 17 years. Because of the decreased malleability and tremendous pressure required to hold the chest wall in the corrected position, post-operative pain control has been a significant problem in this patient population. Thoracic epidurals are commonly employed however mean hospitalizations of up to 7 days have been required before adequate pain control on oral analgesics is obtained and patients are suitable for discharge.

It is hypothesized that using the ON-Q system (I-Flow Corporation, Lake Forest CA) with bilateral intercostal catheter infusion would provide adequate post operative pain control with a significantly shorter hospital length-of-stay than thoracic epidural. Total use of narcotics for 1 week following surgery would also be less with the ON-Q system versus epidural.

DETAILED DESCRIPTION:
Subjects meeting eligibility criteria were randomized to one of two arms for postoperative pain control: the On-Q system versus epidural. All subjects had additional pain management as per standardized protocol including subject controlled intravenous analgesia with morphine equivalent narcotics for a maximum of 48 hours at which time the subject was transitioned to oral pain medications. Subjects using less than 5 mg of Morphine in the first 24 hours after surgery were transitioned to oral pain medications at 24 hours. After transition to oral analgesia, subjects with continued pain assessment greater than 5 were administered intravenous morphine equivalents by nursing staff until pain assessments were less than 5.

ON-Q catheters could have been maintained for up to 6 days. Discharge of subjects with catheters in place was planned. The catheter was removed in the out-patient clinic if the subject was discharged before the 6th day. Subjects with epidural had their epidural discontinued at 72 hours.

Data was recorded for each subject by site personnel while the subjects remained hospitalized, but were recorded in a journal by subjects after discharge up to postoperative day 7.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for repair of their pectus excavatum with minimally invasive (MIRPE) placement of steel or titanium braces at Mayo Clinic Arizona
* Must be able to take oral medications preoperatively and postoperatively.

Exclusion Criteria:

* American Society of Anesthesiology class IV or higher
* Allergic to Ropivacaine or other local anesthetics
* NSAID allergy
* Specific epidural contraindication
* Currently using opioids, sedatives, or hypnotics
* Are pregnant as verified by preoperative pregnancy testing
* Inability to place an epidural, patient refusal for epidural, or failure of an epidural to be properly placed or maintain proper placement for adequate pain control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn E Jaroszewski, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jaroszewski DE, Temkit M, Ewais MM, Luckritz TC, Stearns JD, Craner RC, Gaitan BD, Ramakrishna H, Thunberg CA, Weis RA, Myers KM, Merritt MV, Rosenfeld DM. Randomized trial of epidural vs. subcutaneous catheters for managing pain after modified Nuss in adults. J Thorac Dis. 2016 Aug;8(8):2102-10. doi: 10.21037/jtd.2016.06.62. PMID 27621865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic in Phoenix, Arizona.
Groups:
- ON-Q Soaker Catheter System: ON-Q soaker catheter system with Ropivicaine at 7 cc per hour placed by a single surgeon in the operating room. 7.5" catheters will be tunneled subcutaneously in the anterior axilla bilateral and secured with steri-strips and dressing. ON-Q systems will be primed with 750 cc and refilled accordingly to provide for 6 days of analgesia.
Period: Overall Study
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System
Started | 43 | 42
Completed | 27 | 41
Not Completed | 16 | 1
Not completed — Withdrawal by Subject | 13 | 1
Not completed — Unable to tolerate catheter placement | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for subjects who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System | Total
Number analyzed (Participants) | 27 | 41 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.3 (8.4) | 32.8 (9.4) | 32.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 21 | 31 | 52
Region of Enrollment [Number; unit: participants]
  United States | 27 | 41 | 85

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Hospital length of stay was measured from the day of surgery (day 0) through postoperative day 11.
Time Frame: Up to 11 days post operation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System
Number analyzed (Participants) | 27 | 41
days | 3.5 (0.9) | 3.3 (1.6)
Statistical Analysis 1: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Test type: Superiority or Other; p = 0.55, t-test, 2 sided

2. Primary Outcome: Use of Analgesic Narcotic
Description: Postoperative analgesic used each day over 7 day postoperative period.
Time Frame: 1-7 days post operation
Population: The numbers of participants analyzed varied each day. The numbers per arm analyzed per day category are expressed in the table as (n=Thoracic epidural, ON-Q). The protocol had planned to use the area under the curve, but this was not analyzed in the published paper, due to the presence of missing data in the analgesic narcotic measurements.
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System
Number analyzed (Participants) | 27 | 41
morphine milligram equivalents
  Day 1 (n = 27, 41) | 40.8 (38.5) | 58.7 (45.8)
  Day 2 (n = 27, 41) | 99.5 (71.1) | 107.2 (76.1)
  Day 3 (n = 27, 41) | 79.7 (42.7) | 62.4 (46.9)
  Day 4 (n = 24, 27) | 65.8 (46.1) | 79.4 (57.8)
  Day 5 (n = 12, 13) | 43.5 (33.4) | 78.8 (54.2)
  Day 6 (n = 3, 5) | 30.8 (27.4) | 86.4 (31.9)
  Day 7 (n = 1, 3) | 24.0 (NA) — One participant in the Epidural arm was using an analgesic narcotic on Day 7; a standard deviation cannot be calculated for one participant. | 81.9 (19.0)
Statistical Analysis 1: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between the groups for day 1; Test type: Superiority or Other; p = 0.0872, Unequal Variance T-Test
Statistical Analysis 2: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 2; Test type: Superiority or Other; p = 0.6751, Unequal Variance T-Test
Statistical Analysis 3: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 3; Test type: Superiority or Other; p = 0.1203, Unequal Variance T-Test
Statistical Analysis 4: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 4; Test type: Superiority or Other; p = 0.3582, Unequal Variance T-Test
Statistical Analysis 5: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 5; Test type: Superiority or Other; p = 0.0625, Unequal Variance T-Test
Statistical Analysis 6: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 6; Test type: Superiority or Other; p = 0.0484, Unequal Variance T-Test

3. Secondary Outcome: Mean Daily Pain Score
Description: Pain was measured by a visual analogue scale (VAS) with pre-set markings from 0 to 10, with 0 for no pain to 10 for the worst possible pain. On the case report form each day had 6 time categories: waking up in the morning, around lunch time, afternoon approximately 3-4 pm, dinner time, bedtime, and during the night time. Each day was averaged for each subject, then the values for each arm were averaged.
Time Frame: Days 1-7 post operation
Population: The numbers of participants analyzed varied each day. The numbers per arm analyzed per day category are expressed in the table as (n=Thoracic epidural, ON-Q).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System
Number analyzed (Participants) | 27 | 41
units on a scale
  Day 1 (n = 27, 41) | 2.19 (1.76) | 2.39 (1.72)
  Day 2 (n = 27, 41) | 2.64 (1.41) | 2.60 (1.40)
  Day 3 (n = 27, 41) | 3.16 (1.31) | 2.97 (1.36)
  Day 4 (n = 24, 27) | 3.03 (1.25) | 3.60 (1.19)
  Day 5 (n = 12, 13) | 2.95 (1.22) | 3.30 (1.50)
  Day 6 (n = 3, 5) | 3.28 (0.25) | 3.55 (1.52)
  Day 7 (n=1, 3) | 4.50 (NA) — One participant in the Epidural arm provided a pain score on Day 7; a standard deviation cannot be calculated for one participant. | 4.13 (1.65)
Statistical Analysis 1: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between the groups for day 1; Test type: Superiority or Other; p = 0.6465, Unequal Variance T-Test
Statistical Analysis 2: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 2; Test type: Superiority or Other; p = 0.9233, Unequal Variance T-Test
Statistical Analysis 3: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 3; Test type: Superiority or Other; p = 0.5788, Unequal Variance T-Test
Statistical Analysis 4: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between the groups for day 4; Test type: Superiority or Other; p = 0.1036, Unequal Variance T-Test
Statistical Analysis 5: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 5; Test type: Superiority or Other; p = 0.5314, Unequal Variance T-Test
Statistical Analysis 6: Comparison: Thoracic Epidural vs ON-Q Soaker Catheter System; Comparison between groups for day 6; Test type: Superiority or Other; p = 0.7166, Unequal Variance T-Test

ADVERSE EVENTS:
Time Frame: Adverse event reports were collected from the day of the operation up to postoperative day 7.
Arm/Group | Thoracic Epidural | ON-Q Soaker Catheter System
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/55
Other Adverse Events (participants affected / at risk) | 4/30 | 11/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thoracic Epidural (N=30) | ON-Q Soaker Catheter System (N=55)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pleural effusion requiring thoracentesis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax requiring chest tube (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Urinary retention requiring catheter placement (Renal and urinary disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes